CLINICAL TRIAL: NCT04649177
Title: Pilot Study to Investigate the Feasibility, Reliability and Efficacy of Utilizing OCT to Automate PROSE Fitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Sight (Other)
Collaborators: EYEdeal scanning, LTC (Industry)
Responsible Party: Principal Investigator, Daniel C Brocks, Chief Medical Officer, Boston Sight
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFS-OCT-01
Record Dates: First submitted 2020-11-13; First posted 2020-12-02 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Keratoconus; Ocular Surface Disease; Pellucid Marginal Corneal Degeneration; Ectasia; Corneal Trauma; Corneal Scar; Dry Eye Syndromes; Keratoconjunctivitis Sicca; Sjogren's Syndrome
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic; Corneal Injuries; Dry Eye Syndromes; Keratoconjunctivitis Sicca; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- study group (Other): There is only one study group in this study. All subjects will receive the OCT scanning and PROSE lens fitting.
  Interventions: Device: Ocular surface optical coherence tomography

INTERVENTIONS:
Device: Ocular surface optical coherence tomography — EYEdeal Scanning technology enables rapid measurement of the corneal and scleral topography which provides data for an automated sequence to fit PROSE devices

SUMMARY:
EYEdeal Scanning Technology enables rapid measurement of corneal and scleral topography. By accurately measuring the ocular surface with this imaging technology, the current iterative fitting method required to fit PROSE (prosthetic replacement of the ocular surface ecosystem) devices could be replaced and/or strengthened with a more rapid, automated fitting sequence. This could considerably reduce the time needed per visit, the number of visits, and the number of devices needed to be manufactured to reach the endpoint. Additionally, the scanning technology may afford the opportunity to successfully fit some pathology that were previously treatment failures. The automated technology may as well reduce the intensive clinician training time needed to fit PROSE devices, therefore increasing the availability and access to patients.

The goal of this research is to evaluate the reliability and efficacy of this automated technology for fitting PROSE devices. Data from real-time measurement of the human eye ocular surface topography will be used to fabricate a prosthetic lens. The fit of the PROSE device will be evaluated, as well as the subjective comfort of the fit.

DETAILED DESCRIPTION:
Inclusion and Exclusion Criteria

The participant will be eligible to participate if the following criteria apply:

1. Written Informed Consent has been obtained prior to any study-related procedures
2. Male or female, 18 years of age and older prior to the initial visit
3. Established wearer of PROSE in the study eye with an optimized fit in the opinion of the clinician
4. No medical need for a PROSE retreatment or replacement lens at the time of enrollment in the study eye, in the opinion of the clinician
5. Initial PROSE fitting was initiated and completed at BostonSight, Needham
6. Current PROSE device does not have channels or fenestrations
7. Currently wears a PROSE device in the study eye primarily for an irregular ocular surface /irregular cornea (including but not limited to Keratoconus, Pellucid Marginal Degeneration, Ectasia, Post-Penetrating Keratoplasty, Corneal Scar, Trauma) AND/OR ocular surface disease
8. Has the ability to NOT wear the current PROSE device in the study eye for 3 days prior to scan and 3 days prior to first fitting appointment in the opinion of the investigator and subject
9. In the opinion of the investigator, the subject has the ability to follow study instructions
10. In the opinion of the investigator, the subject has the ability to complete all study procedures and visits

The participant would NOT be eligible to participate if at least one of the following criteria is met:

1. Is currently participating in any other type of eye-related clinical or research study
2. Is pregnant or nursing as reported by the subject
3. Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study
4. Has had previous ocular surgery within the past 12 weeks
5. Intolerance to PROSE wear
6. Inability to maintain stable fixation and exposure for ocular surface imaging
7. Corneal touch by the posterior surface of the device in current PROSE device
8. Allergy to sodium fluorescein
9. Patient is an employee of BostonSight
10. Subject is currently incarcerated.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent has been obtained prior to any study-related procedures
2. Male or female, 18 years of age and older prior to the initial visit
3. Established wearer of PROSE in the study eye with an optimized fit in the opinion of the clinician
4. No medical need for a PROSE retreatment or replacement lens at the time of enrollment in the study eye, in the opinion of the clinician
5. Initial PROSE fitting was initiated and completed at BostonSight, Needham
6. Current PROSE device does not have channels or fenestrations
7. Currently wears a PROSE device in the study eye primarily for an irregular ocular surface /irregular cornea (including but not limited to Keratoconus, Pellucid Marginal Degeneration, Ectasia, Post-Penetrating Keratoplasty, Corneal Scar, Trauma) AND/OR ocular surface disease
8. Has the ability to NOT wear the current PROSE device in the study eye for 3 days prior to scan and 3 days prior to first fitting appointment in the opinion of the investigator and subject
9. In the opinion of the investigator, the subject has the ability to follow study instructions
10. In the opinion of the investigator, the subject has the ability to complete all study procedures and visits

Exclusion Criteria:

1. Is currently participating in any other type of eye-related clinical or research study
2. Is pregnant or nursing as reported by the subject
3. Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study

45. Has had previous ocular surgery within the past 12 weeks

5. Intolerance to PROSE wear

6. Inability to maintain stable fixation and exposure for ocular surface imaging

7. Corneal touch by the posterior surface of the device in current PROSE device

8. Allergy to sodium fluorescein

9. Patient is an employee of BostonSight

10. Subject is currently incarcerated. -

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Brocks, MD, Principal Investigator — Boston Sight
Locations (1):
- BostonSight, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant contributed only one study eye for this study.
Groups:
- Study Group: OCT scanning and PROSE lens fitting based on scan data
Period: Overall Study
Arm/Group | Study Group
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Keratoconus [Count of Participants; unit: Participants] — Keratoconus was determined by slit lamp examination.
  Participants | 10

OUTCOME MEASURES:

1. Primary Outcome: Central Corneal Clearance
Description: Central corneal clearance as measured by OCT after 45 minutes of lens wear Outcome measure reports data only from the study eye.
Time Frame: 45 minutes post lens application
Measure: Mean (Standard Error); unit: microns
Groups:
- Study Group: There is only one study group in this study. All subjects will receive the OCT scanning and PROSE lens fitting based on the scan.
Arm/Group | Study Group
Number analyzed (Participants) | 10
microns | 354.29 (62.68)

2. Primary Outcome: Lens Decentration
Description: Lens decentration after 45 minutes of lens wear (x axis) Outcome measure reports data only from the study eye.
Time Frame: 45 minutes post lens application
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Study Group
Number analyzed (Participants) | 10
microns | 477.89 (190.05)

3. Primary Outcome: Lens Comfort After 45 Minutes of Lens Wear
Description: 0 to 10 grading (0 = very comfortable to 10 = very uncomfortable) Outcome measure reports data only from the study eye.
Time Frame: 45 minutes post lens application
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 10
units on a scale | 2.29 (3.45)

4. Primary Outcome: Number of Participants With Lens Centration
Description: Each study eye (one eye from each participant) was evaluated to determine if the lens was "Centered" (yes) or "Decentered" (no) on the eye after 45 minutes of wear.
  Outcome measure reports data only from the study eye. All participants were reported in this outcome measure.
Time Frame: 45 minutes post lens application
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 10
Participants | 5

5. Primary Outcome: Number of Participants With Aligned Scleral Landing Zone
Description: Each study eye (one eye from each participant) was evaluated to determine if the scleral landing zone was properly aligned on the eye (yes) or not properly aligned on the eye (no) after 45 minutes of wear.
  Outcome measure reports data only from the study eye. All participants were reported in this outcome measure.
Time Frame: 45 minutes post lens application
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 10
Participants | 3

6. Secondary Outcome: Lens Rotation
Description: Lens rotation after 45 minutes of wear. Lens rotation was measured using an embedded program in the iTRACE system. The rotation data with image guided fitting with the OCT system was collected to compare with known experience with non-image guided fitting sets (the traditional fitting process), which typically rotate approximately 20-30 degrees on the eye. A lower number may indicate the manufactured lens more closely approximates the contours of the eye.
  Outcome measure reports data only from the study eye.
Time Frame: 45 minutes post lens application
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Study Group
Number analyzed (Participants) | 10
degrees | 28.83 (24.05)

7. Secondary Outcome: Number of Participants Achieving an Acceptable Fitting Lens
Description: Number of participants achieving an acceptable fitting lens after 45 minutes of lens wear. All participants are reported. Outcome measure reports data only from the study eye.
  Is the fit acceptable for dispensing to the patient (yes) or is the fit NOT acceptable for dispensing to patient (no) as evaluated 45 minutes post lens application.
Time Frame: 45 minutes post lens application
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 10
Participants | 6

8. Secondary Outcome: Number of Participants With Lens Movement
Description: Number of patients with lens movement after 45 minutes of wear are reported. Lens movement (YES) means the lens is NOT appropriately fitting/settling on the eye. Lens movement (NO) means the lens is appropriately fitting/settling on eye. Outcome measure reports data only from the study eye.
Time Frame: 45 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 10
Participants | 4

9. Secondary Outcome: Number of Participants With Adequate Lens Limbal Clearance
Description: Each study eye (one eye from each participant) was evaluated to determine if there was adequate (yes) lens limbal clearance or inadequate (no) lens limbal clearance after 45 minutes of wear.
  Outcome measure reports data only from the study eye. All participants were reported in this outcome measure.
Time Frame: 45 minutes post lens application
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 10
Participants | 7

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04649177/Prot_002.pdf
  • Informed Consent Form (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT04649177/ICF_003.pdf